CLINICAL TRIAL: NCT05072808
Title: Improving Asthma Referrals Following Emergency Department Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Amy Delaroche, Assistant Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB-19-09-1259
Record Dates: First submitted 2021-09-22; First posted 2021-10-11 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Asthma in Children
Keywords: Asthma; Emergency Department; Children; Referral; Pediatric Asthma Control and Communication Instrument for the Emergency Department; PACCI-ED
MeSH Terms: conditions — Asthma; Emergencies

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): ED Providers randomized to the Intervention Group will be able to view the results of the parent-completed questionnaire, the Pediatric Asthma Control and Communication Instrument for the Emergency Department (PACCI-ED), and outpatient referral recommendations aligned with asthma severity.
  Interventions: Other: View PACCI-ED and referral recommendations
- Control Group (No Intervention): ED providers randomized to the Control Group will neither receive the results of the parent-completed PACCI-ED or specific recommendations for outpatient referrals. Patients randomized to the control group will receive usual care.

INTERVENTIONS:
Other: View PACCI-ED and referral recommendations — Results of parent completed PACCI-ED and referral recommendations
  Arms: Intervention Group

SUMMARY:
Asthma is the most common chronic condition among children and many children seek emergency department (ED) care. A key aspect of ED asthma management at the time of discharge is appropriate outpatient referral. Part of the challenge for ED providers is determining which patients require intensive outpatient support as ED providers often do not have the time or familiarity with the asthma guidelines to appropriately stratify asthma severity. Thus, the aim of this study is to determine whether the proportion of children referred to outpatient asthma care can be improved by incorporating a previously validated tool [the Pediatric Asthma Control and Communication Instrument for the Emergency Department (PACCI- ED)] into ED clinical care.

DETAILED DESCRIPTION:
Emergency department (ED) physicians play an important role in the management of pediatric asthma through acute intervention, family education, and appropriate referral to outpatient resources. However, time constraints in the ED limit physicians' ability to appropriately stratify both asthma severity and outpatient referrals. The Pediatric Asthma Control and Communication Instrument for the Emergency Department (PACCI-ED) improves ED providers assessment of asthma control and disease burden. We hypothesize that implementation of the PACCI-ED at the point of care may help to facilitate appropriate referrals to outpatient asthma care.

ED providers will be randomized to the control or intervention group. Providers in the intervention group will receive the results of the parent-completed PACCI-ED accompanied by a one page summary of referral recommendations aligned with asthma guidelines and based upon asthma severity. Providers in the control group will not receive this information and will provide 'usual care'. All providers will complete a brief demographic questionnaire. School-aged children with a history of asthma presenting to the ED for an asthma exacerbation and discharged home who consent to participate will be assigned to the control or the intervention group based upon the ED provider caring for the patient during their ED encounter. Parents will complete a brief demographic questionnaire, the PACCI-ED, and answer two short qualitative audio-recorded questions about barriers to asthma care during their ED visit. Following the ED visit, additional data will be abstracted from the electronic medical record including outpatient referrals placed at the time of ED discharge and follow-up with the referrals within a one-month time-frame.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to Children's Hospital of Michigan (CHM), Detroit, Emergency Department (ED) for an acute asthma exacerbation
* History of asthma as reported by parents

Exclusion Criteria:

* Transfer from outside ED for a higher level of care
* Admitted to the hospital following pediatric ED evaluation
* Significant co-morbidity (pulmonary, cardiac, or other systemic disease)
* Hemodynamic instability
* Non-English speaking
* Previously enrolled in this study
* Patients without their primary caregiver at ED presentation
* Not under the care of CHM ED provider who has consented to be a part of the study

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Proportion of referrals | Eight months
  Proportion of referrals for outpatient asthma care placed in the electronic medical record.

SECONDARY OUTCOMES:
Proportion of subspecialty referrals | Eight months
  Proportion of subspecialty referrals for outpatient asthma care (e.g. allergy/immunology, pulmonology) placed in the electronic medical record.
Patient and provider characteristics | Eight months
  Patient (e.g. age, asthma history) and provider (e.g. training, years in practice) self-reported demographics.
Completed outpatient clinic visits following a referral | 30 days following the ED visit
  Number of patients attending the outpatient clinic visit within 30 days of the referral requested in the electronic medical record at the time of the ED visit.

CONTACTS AND LOCATIONS:
Overall Officials: Amy M DeLaroche, MBBS, Principal Investigator — Detroit Medical Center
Locations (1):
- Children's Hospital of Michigan, Detroit, Michigan, United States

REFERENCES:
- [Background] Akinbami LJ, Moorman JE, Simon AE, Schoendorf KC. Trends in racial disparities for asthma outcomes among children 0 to 17 years, 2001-2010. J Allergy Clin Immunol. 2014 Sep;134(3):547-553.e5. doi: 10.1016/j.jaci.2014.05.037. Epub 2014 Aug 1. PMID 25091437
- [Background] Rachelefsky GS, Kennedy S, Stone A. Enhancing the role of the emergency department in the identification and management of childhood asthma. Pediatrics. 2006 Apr;117(4 Pt 2):S57-62. doi: 10.1542/peds.2005-2000b. No abstract available. PMID 16777838
- [Background] Goldberg EM, Laskowski-Kos U, Wu D, Gutierrez J, Bilderback A, Okelo SO, Garro A. The Pediatric Asthma Control and Communication Instrument for the Emergency Department (PACCI-ED) improves physician assessment of asthma morbidity in pediatric emergency department patients. J Asthma. 2014 Mar;51(2):200-8. doi: 10.3109/02770903.2013.859267. Epub 2013 Dec 4. PMID 24219842
- [Background] Wu DJ, Hipolito E, Bilderback A, Okelo SO, Garro A. Predicting future emergency department visits and hospitalizations for asthma using the Pediatric Asthma Control and Communication Instrument - Emergency Department version (PACCI-ED). J Asthma. 2016;53(4):387-91. doi: 10.3109/02770903.2015.1115520. Epub 2016 Jan 22. PMID 26667853
- [Background] Pade KH, Agnihotri NT, Vangala S, Thompson LR, Wang VJ, Okelo SO. Asthma specialist care preferences among parents of children receiving emergency department care for asthma. J Asthma. 2020 Feb;57(2):188-195. doi: 10.1080/02770903.2019.1565768. Epub 2019 Jan 21. PMID 30663904